CLINICAL TRIAL: NCT02168036
Title: Evaluation of the Mediastinal Lymph Nodes With Endobronchial-Guided Transbronchial Needle Aspiration in Individuals With Lung Diseases
Brief Title: Study of Biologic Materials From the Mediastinal Lymph Nodes From Patients With Lung Disease.
Status: Terminated | Type: Observational
Why Stopped: Study was terminated due to lack of funding.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1104011629
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Lung Disease; Inflammation; Lung Cancer; Sarcoidosis
Keywords: lung disease; mediastinal lymph node; bronchoscopy; Endobronchial-Guided Transbronchial Needle Aspiration
MeSH Terms: conditions — Lung Diseases; Inflammation; Lung Neoplasms; Sarcoidosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Mediastinal tissue/ Lung biological samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with lung disease: General admission criteria for this project will require at least one of the following: (1) symptoms consistent with pulmonary disease with mediastinal lymph node involvement ; (2) chest X-ray and chest CT scan consistent with lung disease and mediastinal lymph node involvement; (3) Individuals with a lung biopsy consistent with lung disease and presenting with enlarged mediastinal lymph nodes; and (4) patients with diseases of organs with known association with lung disease and mediastinal lymph node involvement.

SUMMARY:
The purpose of this protocol is to obtain biologic materials from the mediastinal lymph nodes from patients with lung disease and mediastinal lymph node involvement in order to: (1) develop a better understanding of the cause and development of lung disorders involving the mediastinal lymph nodes; (2) identify biologic parameters that help diagnose and predict the behavior of human lung diseases; and (3) identify individuals who will be suitable candidates for other protocols such as those involving investigational new drugs.

DETAILED DESCRIPTION:
This study will use bronchoscopy with endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) as part of their diagnostic work up as recommended by the treating physician. The procedure will be performed as standard of care, either under general anesthesia in the operating room or in the bronchoscopy suite under moderate sedation and analgesia. Bronchoscopy with EBUS-TBNA is normally an ambulatory procedure. During the procedure, biopsy needle will be passed through the tube and a small sample will be taken for both diagnostic and research purposes. Samples collected for diagnostic purposes will be sent to the Department of Pathology. Additional biopsy samples will be collected for research purposes. The subject is observed after the bronchoscopy, including vital signs and level of consciousness, until they are back to baseline. All subjects will be discharged with an escort as per Hospital policy. An overnight stay would be required for ambulatory individuals only if the individual is not, in the judgment of the treating attending physician, safe to be discharged as is standard practice.

ELIGIBILITY:
Inclusion Criteria:

* Must provide informed consent
* Males and females, age 18 years and older
* Lung disease proven by at least one of the following:

  1. symptoms consistent with pulmonary disease
  2. chest X-ray and chest CT and/or PET CT scan consistent with lung disease and mediastinal lymph node involvement
  3. lung biopsy consistent with lung disease known to involve mediastinal lymph nodes
  4. patients with diseases of organs with known association to lung disease and mediastinal lymph node involvement.
* Undergoing fiberoptic bronchoscopy with EBUS-TBNA as dictated by their standard clinical care

Exclusion Criteria:

* Patient refuses consent.
* Any history of allergies to xylocaine, lidocaine, versed, valium, atropine, or any local anesthetic will not be included in the study
* Individuals who cannot tolerate general anesthesia or moderate sedation and analgesia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diseases of organs with known association with lung disease and mediastinal lymph node involvement.
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2011-08-16 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-16 (Actual)

PRIMARY OUTCOMES:
Evidence that is consistent with lung disease and presentation of enlarged mediastinal lymph nodes | 24 Hours
  Bronchoscopy with endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA)

CONTACTS AND LOCATIONS:
Overall Officials: Ben-Gary Harvey, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College and Weill Cornell Medical Center, Department of Genetic Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided